CLINICAL TRIAL: NCT07125053
Title: Optimizing Effectiveness and Implementation of COPD Self-Management Treatment
Brief Title: COPD Resources, Education, and Activity Designed for You Study
Acronym: COPD READY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Chicago (Other); American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ORA# 23050802; R01HL173120-01A1 (NIH)
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: COPD
Keywords: copd; emphysema; chronic bronchitis; self-management; lifestyle management; physical activity; inhaler use; patient education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Motor Activity | interventions — Educational Status; Exercise

STUDY DESIGN:
Intervention Model Description: 2x2x2 factorial study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition #1 (Experimental): Education = self-guided; Physical Activity = on; Inhaler Training = on
  Interventions: Behavioral: Education (self-guided); Behavioral: Physical Activity; Behavioral: Inhaler Training
- Condition #2 (Experimental): Education = self-guided; Physical Activity = on; Inhaler Training = off
  Interventions: Behavioral: Education (self-guided); Behavioral: Physical Activity
- Condition #3 (Experimental): Education = self-guided; Physical Activity = off; Inhaler Training = on
  Interventions: Behavioral: Education (self-guided); Behavioral: Inhaler Training
- Condition #4 (Experimental): Education = self-guided; Physical Activity = off; Inhaler Training = off
  Interventions: Behavioral: Education (self-guided)
- Condition #5 (Experimental): Education = counselor-led; Physical Activity = on; Inhaler Training = on
  Interventions: Behavioral: Education (counselor-led); Behavioral: Physical Activity; Behavioral: Inhaler Training
- Condition #6 (Experimental): Education = counselor-led; Physical Activity = on; Inhaler Training = off
  Interventions: Behavioral: Education (counselor-led); Behavioral: Physical Activity
- Condition #7 (Experimental): Education = counselor-led; Physical Activity = off; Inhaler Training = on
  Interventions: Behavioral: Education (counselor-led); Behavioral: Inhaler Training
- Condition #8 (Experimental): Education = counselor-led; Physical Activity = off; Inhaler Training = off
  Interventions: Behavioral: Education (counselor-led)

INTERVENTIONS:
Behavioral: Education (self-guided) — The self-guided eduction program consists of a mailed booklet entitled, "Learning to live with COPD," along with two additional mailings with information on the ALA's Patient and Caregiver Network and the Respiratory Health Association's COPD Caregiver's Toolkit.
  Arms: Condition #1; Condition #2; Condition #3; Condition #4
Behavioral: Education (counselor-led) — The counselor-led education program combines mailings with phone counseling delivered by ALA Lung Helpline counselors. Three phone sessions (20-30 minutes each) are completed over the course of 6 weeks in the main treatment phase, with two additional optional booster sessions offered between 6 and 12-weeks post-randomization. The counselor-led program follows a structured outline of curriculum for each session, focusing on the topic areas of developing a COPD exacerbation action plan, recognizing COPD exacerbations, and coping with breathlessness.
  Arms: Condition #5; Condition #6; Condition #7; Condition #8
Behavioral: Physical Activity — The physical activity program will consist of a personalized prescription for home-based exercise following published guidelines, consisting of aerobic, strengthening, and flexibility exercises, tailored to participants' current fitness level and dyspnea symptoms. Aerobic exercise will incorporate ground-based walking training, a well-established, safe, and feasible physical activity program for individuals with COPD. Participants will complete three videoconference sessions (30-45 minutes each) over the course of 6 weeks in the main treatment phase, with two additional optional booster sessions between week 6 and 12.
  Arms: Condition #1; Condition #2; Condition #5; Condition #6
Behavioral: Inhaler Training — Participants will receive inhaler technique education using a virtual teach-to-goal method. In each session, individuals are observed using their inhaler, provided feedback, and then observed again. Inhaler technique is scored using a checklist specific to each inhaler device. Participants will complete two inhaler training sessions via videoconference at week 1 and week 4, with an optional booster session offered at week 8.
  Arms: Condition #1; Condition #3; Condition #5; Condition #7

SUMMARY:
Although COPD self-management treatment programs are effective in reducing COPD-related hospitalizations and increasing quality of life, there is a limited understanding of 'how and why' they work. The proposed research will use an engineering-inspired study design to identify effective COPD self-management treatment components and guide its 'real world' implementation. The long-term goal of this line of research is to build an optimized COPD self-management program, and scale the program up to reduce the burden of COPD at a population health level.

DETAILED DESCRIPTION:
The study's overall objective is to test component effects of COPD self-management treatment and select an optimized treatment program, while simultaneously gathering information on factors impacting implementation (i.e., Hybrid Type 1 Effectiveness-Implementation Study).1 The study design is guided by the Multiphase Optimization Strategy (MOST),2 an innovative, engineering-inspired methodological framework for intervention development that uses highly efficient randomized experimentation to assess the performance of treatment components on clinically-relevant outcomes, independently and in combination. The proposed research will achieve the following Specific Aims:

Aim 1. Determine the main and interactive effects of three treatment components (i.e., self-management education, inhaler training, and physical activity) on a) respiratory-related hospitalizations over 12 months (primary outcome), and b) health-related quality of life (secondary outcome) by conducting a 2x2x2 factorial experiment. Program costs associated with delivery of each treatment condition will be measured and mediation analyses will be conducted to further understand the mechanisms of component effects.

Sub-Aim 1a. Examine the interaction of baseline disease severity and comorbid conditions (i.e., cardiovascular disease, lung cancer, sleep apnea, metabolic syndrome) with each treatment component on outcomes, to explore potential differences in treatment response.

Aim 2. Select the optimized treatment program. The investigators will identify the optimized treatment package that produces the best expected outcomes (i.e., reduction in respiratory-related hospitalizations and increased health-related quality of life), while maintaining efficiency in the program cost for treatment delivery.

Aim 3. Develop a set of implementation strategies to increase referrals to the optimized treatment program by conducting a mixed methods process evaluation with healthcare providers (N=10-20) and administrators (N=10-20). Informed by the Consolidated Framework for Implementation Research (CFIR), the investigators will assess the barriers and facilitators impacting the program referral workflow, and use this data to inform selection of implementation strategies to increase referrals.

ELIGIBILITY:
Inclusion Criteria:

* Residence in the continental United States
* Age 40 years or older
* Report a physician diagnosis of COPD
* Report a COPD-related hospitalization over the past 12 months
* Use an inhaled medication for COPD at least once per week
* Have access to a connected device (i.e., smartphone, tablet, and/ or computer) to complete study procedures

Exclusion Criteria:

* COPD exacerbation within the past month
* New or worsening chest pain that happens without exertion
* Cognitive dysfunction impairing ability to provide informed consent and follow study procedures
* Terminal illness (i.e., < 6 month life expectancy) that is non-COPD related
* Living at a chronic care facility (i.e., nursing home, assisted living)
* Inability to participate in mild physical activity such as walking, stretching, and lower limb exercises
* Inability to speak/ read English

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
12-month respiratory-related hospitalization | 12 months
  Incidence of one or more respiratory-related hospitalization at 12-month follow-up

SECONDARY OUTCOMES:
Health-related quality of life | 12 weeks
  Change in Chronic Respiratory Disease Questionnaire (CRQ)-Mastery subscale score from baseline to 12-week follow-up. A mean score will be computed for the CRQ-Mastery subscale (range 1-7), with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R. Mathew, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographics, social determinants of health, clinical trial results, medical records, audio recordings, and survey/ questionnaire data will be collected from a total of 448 adult participants in a nationwide study. Our intent is to share research data to the greatest extent possible, and there are only a few considerations that require us to limit the type and amount of data shared. Given the potential to deduce participant identities from a combination of geographic location and demographic factors, we will not be share geographic data (e.g., Census tract identifiers) or any data extracted from publicly available databases based on participant's residential address. Any intellectual property resulting from this study that can be patented will remain easily and widely available to the researchers in accordance with the NIH Principles and Guidelines. Distribution of resources to for-profit entities may occur under material transfer agreements or non-exclusive license arrangements.
Supporting Information: Study Protocol
Time Frame: Data will be made available as soon as possible after the data collection period has ended and will occur no later than the end of the project period or the time of any publication after the study investigators have had reasonable time to prepare manuscripts. Data will remain available for a period of at least 10 years. (i.e., 9/1/29-9/1/39).
Access Criteria: Access to the data generated through this project will be granted upon review of a brief request form, completed by the requesting party, that summarizes the intended use of the data (e.g., the nature of any planned analyses), their qualifications, their institutional affiliation, and any required regulatory approval for the planned work by their IRB or other regulatory body. Data sharing will conform to any restrictions specified by regulatory bodies, such as IRBs and institutional Privacy Offices. A Data Use Agreement may be required, depending on the nature of the data requested, at the discretion of our institution's IRB, Office of Legal Affairs, or Privacy Office. Our plan is to deposit research data in the Open Science Framework data archive, an established, publicly accessible repository with a multitude of advantageous features.